CLINICAL TRIAL: NCT05178849
Title: QUALHYBOM : Therapeutic Communication Associated With Local Anesthesia Versus Local Anesthesia During Bone Marrow Biopsy: Clinical, Controlled, Randomized, Multicenter Study
Brief Title: QUALHYBOM Hypnosis Versus Equimolar Mixture of Oxygen and Nitrous Oxide (MEOPA) During a Bone Marrow Biopsy: a Clinical, Controlled, Randomized, Multicenter Study
Acronym: QUALHYBOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC19_8879_QUALHYBOM; IDRCB (Other: 2023-A00039-36); SI RIPH2G (Other: 23.00615.000256)
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Bone Marrow Biopsy
Keywords: Hypnosis
MeSH Terms: interventions — Hypnosis; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized, single-blind, multicenter study comparing two approaches to analgesia during BOM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis + local anesthasia (Experimental): As part of this project, local anesthesia will be supported by hypnosis in patients randomized to the "hypnosis + AL" arm, and started as soon as the patient is in prone position.
  Hypnosis is a particular psychological state marked by the functioning of the individual at a level of attention other than the ordinary state of consciousness. It can, under certain conditions, give the appearance of sleep or sleepwalking without sharing all of its characteristics.
  As part of care, hypnosis is widely used for pain control. The side effects reported are nil. One of its main benefits is improved patient comfort. One of its main benefits is improved patient comfort.
  For the local anesthesic, the doctor uses in both arms of the study a 20 ml vial of lidocaine hydrochloride without adrenaline for injection dosed at 2%.
  Interventions: Other: Hypnosis; Drug: Local anesthetic
- Local anesthesia (Active Comparator): For the local anesthesic, the doctor uses in both arms of the study a 20 ml vial of lidocaine hydrochloride without adrenaline for injection dosed at 2%.
  Interventions: Drug: Local anesthetic

INTERVENTIONS:
Other: Hypnosis — Hypnosis
  Arms: Hypnosis + local anesthasia
Drug: Local anesthetic — For the local anesthesic, the doctor uses in both arms of the study a 20 ml vial of lidocaine hydrochloride without adrenaline for injection dosed at 2%.

SUMMARY:
The Osteo-Medullary Biopsy (BOM) is a procedure carried out by means of a trocar and makes it possible to obtain a bone core. This gesture is usually performed by performing a local subcutaneous anesthesia at the puncture point of the postero-superior iliac crest, sometimes associated with the use of MEOPA (equimolar mixture of oxygen and nitrous oxide) in case of persistence a painful perception at the puncture site during the examination, in accordance with the Guide to Good Practices for Spinal Puncture of the French Society of Hematology. However, this procedure appeared to us to be insufficient to ensure optimal comfort and effective analgesia and to effectively control anxiety. The realization of the BOM under hypnosis represents an alternative which can bring additional comfort to the patient thanks to a better tolerance and a reduction in the perception of pain. During hypnosis, it has been demonstrated that the stimulation of cortical areas in sleep and in wakefulness leads to a reduction in the pain felt by the patient. Thanks to a retrospective study carried out within the hematology department of the University Hospital of Rennes, we observed a net benefit of hypnosis on the comfort and the pain felt during the realization of a bone marrow biopsy, associated with a decrease in anxiety. In addition, the number of cubicles obtained during the examination (proportional to the size of the biopsy core) was better. Obtaining more than 10 cubicles (figure required by pathologists for a quality examination) was observed in 78% of cases with hypnotic support versus 53% without hypnotic support. Finally, the sample-taking physician reported better operational comfort when accompanied by the hypnotherapist nurse.

DETAILED DESCRIPTION:
This original project aims, on the one hand, to improve the conditions for carrying out a procedure known to be invasive and painful and, on the other hand, to ensure better quality. So far, only one randomized study has been reported on the use of hypnosis in adults during a bone marrow biopsy showing a significant improvement in the anxiety generated by this test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Naive patient of BOM;
* Support at the day hospital;
* Affiliated with a social security scheme;
* Having signed a free, informed and written consent.

Exclusion Criteria:

* Patients requesting that the BOM be performed under MEOPA;
* Pregnant or breastfeeding woman;
* Emergency surgery;
* Patients consuming long-term opiates preoperatively;
* Substance addiction ;
* Patient unable to understand the rating scales;
* Palliative care patients;
* Deaf and / or dumb patients;
* Patients with psychiatric pathologies (schizophrenia, bipolarity);
* Adult persons subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Comfort | 3 minutes (+/- 1 minute) after the end of the gesture, or just before MEOPA administration if applicable
  Patient comfort will be assessed by a simple, validated digital comfort scale. This scale is graduated from "0" (no comfort) to "10" (maximum conceivable comfort). This evaluation will be carried out 3 minutes (+/- 1 minute) after the end of the gesture.

SECONDARY OUTCOMES:
Pain visual analogue scale | Immediately after the assessment of the comfort scale
  The patient's pain will be assessed by the visual analogue scale (VAS). This scale is graduated from "0" (no pain) to "10" (maximum pain imaginable). It will be performed immediately after the assessment of the comfort scale.
Anxiety | 10 minutes (+/- 3 minutes) before the biopsy procedure and repeated immediately after the biopsy procedure (just after the pain assessment)
  The anxiety felt by the patient will be assessed by a simple and validated numerical scale. This scale is graduated from "0" (no anxiety) to "10" (maximum anxiety imaginable). It will be performed 10 minutes (+/- 3 minutes) before the biopsy procedure and repeated after the biopsy procedure (just after the pain assessment).
Practitioner's comfort | Immediately after leaving the patient's room
  The comfort of the practitioner during the taking of the sample will be evaluated by the simple and validated digital comfort scale. This scale is graduated from "0" (no comfort) to "10" (maximum conceivable comfort). This assessment will be performed by IDE-H immediately after leaving the patient's room.
Number of stalls | 1 day (At BOM's gesture)
  The quality of the sample will be assessed by the pathology laboratory according to the number of stalls present on the biopsy: biopsies ≥ 10 stalls will be considered of sufficient quality while biopsies <10 stalls will be deemed of insufficient quality.
MEOPA administration | Through gesture completion, an average of 45 minuts
  MEOPA administration or not during the gesture

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Vannes hospital, Vannes, Britanny
  - Rennes University Hospital, Rennes, Brittany Region
  - Orléans Hospital, Orléans
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No